CLINICAL TRIAL: NCT04157491
Title: A Single-center, Single-arm, Phase II Trial to Evaluate the Efficacy and Safety of Anti-PD-1 Antibody Combined With Anlotinib in the Treatment of Recurrent or Advanced Endometrial Cancer
Brief Title: Anti-PD-1 Antibody Combined With Anlotinib in the Treatment of Endometrial Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jundong Li, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SINAL1618
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; anlotinib; anti PD-1 antibody
MeSH Terms: conditions — Endometrial Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib and anti PD-1 antibody (Experimental)
  Interventions: Drug: anlotinib and anti PD-1 antibody

INTERVENTIONS:
Drug: anlotinib and anti PD-1 antibody — Anti-PD-1 antibody administered by intravenous (IV) infusion on Day 1 of each 21-day cycle plus Anlotinib 12 mg administered orally (PO) once daily (QD) Day1-Day14 during each 21-day cycle.

SUMMARY:
The purpose of the study is to evaluate the Efficacy and safety of Anti-PD-1 antibody combined With anlotinib in the treatment of recurrent or advanced endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age and female;
2. Histologically confirmed diagnosis of endometrial cancer；
3. Patients must have received at least 1 cycle of platinum-based chemotherapy；

   * Patients with recurrent endometrial cancer that has failed at least one line of platinum-based system chemotherapy
   * Patients with newly diagnosed advanced endometrial cancer has persist lesion after standard treatment with surgery and chemotherapy ± radiotherapy （at least one line of platinum-based systemic chemotherapy）
4. At least one measurable lesion according to RECIST1.1 on CT;
5. ECOG performance status 0-2;
6. Life expectancy ≥ 3 months;
7. Adequate hepatic, renal, heart, and hematologic functions. Absolute Neutrophil Count(ANC) ≥ 1.5×109/L, Platelet (PLT) ≥ 70×109/L, Hemoglobin(HGB) ≥ 80 g/L, total bilirubin within 1.5×the upper limit of normal (ULN), and serum transaminase≤2.5×Upper Limit Of Normal(ULN), serum creatine ≤ 1.5 x Upper Limit Of Normal(ULN), creatinine clearance rate ≥50ml/min, International Normalized Ratio<1.5 x Upper Limit Of Normal(ULN), Urinary protein≤（+）and Thyroid stimulating hormone≤ 1.5 x Upper Limit Of Normal(ULN).
8. Signed and dated informed consent.

Exclusion Criteria:

1. Pathology confirmed with sarcoma components (including malignant mixed mullerian tumors, endometrial leiomyosarcoma, and endometrial stromal sarcoma);
2. Exposured to any anti-tumor drugs within 4 weeks;
3. Less than 4 weeks since the patient underwent any major surgery or expect a major surgery during trial;
4. Radiation therapy within 21 days（Palliative radiotherapy for bone metastases within14 days）;
5. Exposured to any anti-PD1 antibody drugs；
6. Any unresolved toxicity CTCAE > Grade 1 from the prior chemoradiation therapy（Excluding hair loss and neurotoxicity）;
7. Current or prior use of any immunosuppressive medication or systemic hormone therapy（which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid Prednisone>10mg/d）within 14 days before the first dose of anti-PD1 antibody and Anlotinib；
8. Any primary malignancy within 5 years (except for fully treated in situ malignant such as breast cancer, bladder cancer, cervical carcinoma in situ, cutaneous basal cell carcinoma or squamous cell carcinoma);
9. History of psychiatric drugs abuse and not be abstinent, or dysphrenia；
10. Central nervous system diseases, including uncontrollable epilepsy and symptomatic brain metastases;
11. Digestive diseases that may affect drug absorption (such as atrophic gastritis)
12. Active ulcers, intestinal perforation, intractable intestinal obstruction, and history of digestive tract perforation within 28 days prior to enrollment；
13. Uncontrolled hypertension（blood pressure >140/90 mmHg after adequate treatment）;
14. Severe cardiovascular disease: unstable angina pectoris, myocardial infarction, grade III-IV cardiac insufficiency (NYHA standard), and peripheral vascular disease above 2 degrees within 6 months prior to enrollment;
15. Severe arrhythmia requiring drug control, QT interval >470ms；
16. Active hemorrhage or hemorrhage tendency.
17. Within 6 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack (TIA), hematencephalon, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc.
18. Active infections such as HIV/AIDS or other serious infectious diseases
19. Any active autoimmune disease or history of autoimmune disease (including but not limit to autoimmune hepatitis, interstitial pneumonia, hepatitis, enteritis, nephritis, hyperthyroidism, pituitary inflammation, vasculitis, uveitis) . Patients need receiving systemic hormonal therapy and/or immunosuppressive therapy (eg asthma requiring bronchodilators);
20. Receipt of live attenuated vaccination within 30 days prior to study entry;
21. Known to be allergic to any drug in the study;
22. For women of child-bearing age, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative. They will take appropriate methods for contraception during the study.
23. Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | Approximately 24 months.
  Objective tumor response was defined as the proportion of patients whose tumor volume has been reduced to a predetermined value and can be maintained for more than 4 weeks, ie ORR=CR+PR.

SECONDARY OUTCOMES:
Duration of Response(DoR) | Approximately 24 months.
  Duration of response was defined as the time when the tumor is first evaluated as CR or PR to the first assessment for PD or for any cause of death.
Disease Control Rate(DCR) | Approximately 24 months.
  Disease control rate was defined as the proportion of subjects with complete response (CR) or partial response (PR) or disease stabilization (SD) in the analyzed population according to the RECIST 1.1 criteria.
Time to Objective Response(TTR) | Approximately 24 months.
  Time to objective response was defined as the time from the start of treatment to the first objective tumor remission (CR or PR).
Progression Free Survival(PFS) | Approximately 24 months.
  Progression-free survival was defined as the duration of time from study entry to time of progression, death, or the date of last contact, whichever occurs first.
Overall Survival（OS） | Approximately 48 months.
  Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Overall Survival Rate at 12 months | Approximately 12 months.
  Overall survival rate at 12 months was defined as the proportion of patients who were still alive in 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wei W, Ban X, Yang F, Li J, Cheng X, Zhang R, Huang X, Huang Y, Li Q, Qiu Y, Zheng M, Zhu X, Li J. Phase II trial of efficacy, safety and biomarker analysis of sintilimab plus anlotinib for patients with recurrent or advanced endometrial cancer. J Immunother Cancer. 2022 May;10(5):e004338. doi: 10.1136/jitc-2021-004338. PMID 35623659